CLINICAL TRIAL: NCT07090590
Title: Evaluating Feasibility, Acceptability, Usability, and an Initial Estimate of Effect of a Novel Training Platform on Peer Recovery Supporter Skill, Adherence, and Knowledge Gain
Brief Title: Evaluating Feasibility, Acceptability, Usability, and an Initial Estimate of Effect of a Novel Training Platform on Peer Recovery Supporter Skill, Adherence, and Knowledge Gain-Phase I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thrive Digital Health, LLC (Industry)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 4R44AA030953-Phase I; 1R44AA030953-01A1 (NIH)
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Substance-related Disorders; Alcohol and Other Substance Use Prevention; Alcohol and Other Drug Use Disorders
Keywords: Peer Recovery Support; Peer Recovery Coaching; Substance Use Recovery; Alcohol Use Disorder
MeSH Terms: conditions — Substance-Related Disorders; Alcoholism

STUDY DESIGN:
Intervention Model Description: feasibility/usability pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TDPP Training Intervention (Experimental): Participants in this arm received access to the Thrive Digital Peer Platform (TDPP), a fully asynchronous, self-paced digital training program designed to build skills in Peer Recovery Support Specialists (PRSS). The TDPP includes 11 interactive modules structured around the Connect, Grow, Apply (CGA) learning model, peer-led stories, scenario-based exercises, and knowledge assessments. No control or comparator arm was included.
  Interventions: Behavioral: Thrive Digital Peer Platform (TDPP)

INTERVENTIONS:
Behavioral: Thrive Digital Peer Platform (TDPP) — The Thrive Digital Peer Platform (TDPP) is a fully asynchronous, web-based training program designed to support the professional development of Peer Recovery Support Specialists (PRSS). The platform includes 11 interactive modules structured around the Connect, Grow, Apply (CGA) learning model. Content includes peer-led stories, behavioral simulations, scenario-based learning, and formative assessments. The intervention is intended to build competencies in professionalism, communication, and application of recovery-oriented peer support principles.
  Other Names: TDPP

SUMMARY:
This pilot study evaluates the feasibility, usability, and acceptability of the Thrive Digital Peer Platform (TDPP), an online training system for Peer Recovery Support Specialists (PRSS). Twelve participants were enrolled to complete the full TDPP asynchronous curriculum, including self-paced modules, peer-led storytelling, and applied practice activities. The study aimed to assess participant engagement, satisfaction, and perceived relevance of the training to their work as peer supporters. This work represents the Phase I portion of a Fast Track SBIR funded by the National Institute on Alcohol Abuse and Alcoholism (NIAAA).

DETAILED DESCRIPTION:
The Thrive Digital Peer Platform (TDPP) was developed to support the professionalization and skill development of Peer Recovery Support Specialists (PRSS) by providing an accessible, modular, and evidence-informed training experience. In this Phase I pilot, twelve PRSS participants were recruited to complete a series of interactive online learning modules aligned with the "Connect, Grow, Apply" (CGA) educational framework. Each module contained peer-led narratives, knowledge checks, and behavioral exercises grounded in real-world coaching scenarios.

Primary outcomes included system usability, satisfaction, and self-reported training relevance. Participants completed a post-training assessment and a brief exit interview to capture usability and acceptability ratings. The findings were used to refine content, improve onboarding, and establish readiness for a larger randomized controlled trial in Phase II.

This study did not include a control group. All participants received access to the full training experience and completed their participation within a defined study period. No follow-up or long-term monitoring was conducted.

This trial was conducted as the Phase I component of a Fast Track SBIR (R44AA030953) funded by the National Institute on Alcohol Abuse and Alcoholism (NIAAA).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Self-identified person in recovery from a substance use disorder
* At least one year of continuous sobriety from alcohol and other substances
* Currently working or preparing to work as a Peer Recovery Support Specialist (PRSS)
* Willing and able to participate in digital training sessions
* Has access to a computer, tablet, or smartphone with internet connection
* Able to read and understand English
* Provides informed consent

Exclusion Criteria:

* Active suicidal ideation (as indicated by PHQ-9 item 9)
* An inability to read or speak English
* Severe anxiety (GAD-7 score >15)
* Inability to complete online training due to technical or cognitive limitations

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-03-18 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Skill and Adherence (YACS II) | From baseline to within 1 week after training completion
  Scored performance on videotaped role-play using a modified version of the Yale Adherence and Competence Scale II (YACS II).

SECONDARY OUTCOMES:
System Usability Scale (SUS) Score | Immediately post-training
  Self-reported usability score using the System Usability Scale (SUS), a validated 10-item instrument that assesses the ease of use, satisfaction, and user experience of the TDPP platform.
Knowledge Gain (Pre/Post Assessment) | From baseline to immediately post-training
  Improvement in participant scores on a knowledge test derived from the PRSS curriculum, administered pre- and post-training.
Intention to Use (UTAUT-2 scale) | Immediately post-training
  Assessed using the UTAUT-2 "Intention to Use" construct, scored on a 5-point Likert scale. Measures perceived likelihood of future platform use in practice.

OTHER OUTCOMES:
Self-Reported Satisfaction | Immediately post-training
  Participant-reported satisfaction with the training experience, assessed via a Likert-scale item ("How satisfied were you with the training experience overall?"). Scores range from 1 (not satisfied) to 5 (very satisfied).
Qualitative Feedback (Open-Ended Exit Interview) | Immediately post-training
  Participant reflections on their training experience, collected through a structured exit interview or open-text response field. Thematic content analysis will be used to identify emergent themes related to learning impact, perceived professionalism, and platform usability.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Pesce, JD, MBA, Principal Investigator — Thrive Digital Health
Locations (1):
- Thrive Digital Health, Solon, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
This is a small, single-arm pilot study focused on usability, feasibility, and early-stage training outcomes. No individual participant data will be shared due to the limited sample size, qualitative nature of feedback, and privacy considerations. Aggregate findings may be shared in scientific presentations or publications.